CLINICAL TRIAL: NCT00863044
Title: Impact of High Frequency Ventilation During Coronary Anastomosis in Off Pump Coronary Artery Bypass.
Brief Title: High Frequency Ventilation During Off Pump Coronary Artery Bypass Graft (CABG)
Acronym: VHF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Alain Deschamps, MD, PhD, FRCPC, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-1032
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Coronary Artery Bypass Graft
Keywords: off pump coronary bypass; high frequency ventilation; cerebral oxygen saturation; vasopressors used; right and left ventricular function; arterial blood pressure; heart rate
MeSH Terms: interventions — N(6)-2-(4-aminophenyl)ethyladenosine; High-Frequency Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High frequency ventilation (Active Comparator): high frequency ventilation
  Interventions: Procedure: High frequency ventilation
- Apnea (Placebo Comparator): lung ventilation will be stopped during distal anastomosis as is commonly done
  Interventions: Procedure: Apnea

INTERVENTIONS:
Procedure: Apnea — Ventilation will be stopped for the duration of the anastomosis as it's done currently. At all other times during the surgery, the ventilatory parameters will be adjusted to maintain a PaCO2 between 40 and 45 mmHg.
  Other Names: apnea during anastomosis in off pump CABG
  Arms: Apnea
Procedure: High frequency ventilation — The patients will be ventilated using a tidal volume of 1.5 ml per Kg and a respiratory rate of 100 per minute for as long as the surgeon needs to perform the distal anastomosis of the coronaries.
  Arms: High frequency ventilation

SUMMARY:
This study is to test the safety of high frequency-low volume ventilation during off pump coronary artery bypass as reflected in the near infrared spectroscopy values for cerebral oxygenation.

DETAILED DESCRIPTION:
Ventilatory protocol: Patients will be randomized to either the apnea group or the HFV group. In the HFV group the patients will be ventilated using a tidal volume of 1.5 ml per kg and a respiratory rate of 100 per minute for as long as the surgeon needs to perform the distal anastomosis of the coronaries.The same surgeon will perform all surgeries. In the Control group, ventilation will be stopped for the duration of the anastomosis as it's done currently. At all other times during the surgery, the ventilatory parameters will be adjusted to maintain a PaCO2 between 40 and 45 mmHg.

The anesthesia protocol for the off pump coronary artery bypass will be as follows: premedication will be left at the discretion of the anesthesiologist. In the operating room, the patient will be instrumented with a radial arterial line before induction. Induction will consist of a bolus of 1.0 mcg per Kg of Sufentanil. Anesthesia will be maintained with 1mcg per Kg per hour of Sufentanil. One per cent Isoflurane will be used as hemodynamic parameters allow. Rocuronium 0.7 mg per Kg will be used to facilitate endotracheal intubation. Following endotracheal intubation the patients will monitored with a pulmonary artery catheter and a femoral arterial line. A perfusionist will be on standby at all times for possible conversion to extracorporeal circulation.

Measures to effect:

Routine baseline laboratory investigations will be performed at admission of the patient to the ward.

Hemodynamic parameters:

Arterial blood pressure, heart rate, pulmonary artery pressure, right ventricular pressure will be recorded five minutes intervals throughout the surgery.

Ventilatory parameters and blood gases:

End tidal CO2 and pulse oxymetry will be recorded at five minutes intervals throughout the surgery.

Arterial blood gases will be performed after induction, before and after each distal coronary anastomosis and when judged necessary. The type and time for each anastomosis will be noted.

C-reactive protein and brain natriuretic peptide:

Measurements of CRP and BNP will be perform at admission, after induction of anesthesia, in the intensive care unit after the surgery and 24 hrs after admission to the intensive care unit.

We will use the serum for measure of CRP.CRP will be measured using the Dade Behring N High Sensitivity CRP assay (Dade Behring Diagnostics,Marburg,Germany) on the BN ProSpec Nephelometer (Dade Behring Diagnostics).The assay will use monoclonal anti-CRP antibodies coated to polystyrene particles and a human calibrator traceable to the WHO reference material. We will use the Heparinised Plasma for measure of NT Pro-BNP.NT Pro-BNP will be measure by electrochemiluminescence immunoassay using the Roche Pro BNP assay (Roche Diagnostics , Mannheim,Germany) on the ElecSys 2010 analyzer (Roche Diagnostics).This assay will use two polyclonal antibodies in a sandwich format.

Cerebral Oximetry Monitoring:

Cerebral oxymetry (rSO2) using near infrared spectroscopy (NIRS, Invos 5100; Somanetics Corporation, Troy, MI) will be performed on all patients. After cleaning adjacent skin area with alcohol, an adhesive optode pad will be placed over each front-temporal area. Resting baseline rSO2 values will be obtained after waiting at least 1 min after placement of sensors once values had stabilized, with patient resting quietly and receiving 3-5 L of O2/min by nasal cannula. Continuous rSO2 values will be store on a floppy disk with a 15 s update for the duration of the intraoperative period. With application of the chest dressing, and before leaving the OR, monitoring will be discontinued and optodes will be removed.

Transesophageal echocardiographic (TEE) measurements:

A comprehensive TEE examination will be performed for all patients as it's done routinely(25). Specific TEE measurements as recommended be the ASE will be perform before and after distal coronary anastomosis(26). RVMPI will be defined as the sum of isovolumic contraction time and isovolumic relaxation time divided by the ejection time and the normal value is 0.28±0.04). RV MPI will be measured using both pulse wave and tissue Doppler imaging from a deep transgastric view and upper esophageal view. Right ventricular FAC % will be measure in 4 chambers view and calculated as RV change in area in diastole minus RV change in area in Systole divided by the calculated RV area in Diastole (37).

Analysis of HR and BP variability:

Baseline HR and BP variability will be analysed using wavelet transformation (27). The extraction of characteristic frequencies, or specific oscillations, of a signal that is composed of the consecutive R-R intervals for HR variability analysis, or consecutive systolic blood pressures for BP variability analysis, is used. The analysis will be made using MATLAB® and the dedicated toolbox software Wavelab. High frequency power of the HR variability is indicative of changes in parasympathetic nervous system. Total power of the BP variability signal is used as a measure of sympathetic outflow.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Patients able to give consent with knowledge of french or english language.

Exclusion Criteria:

* Patients undergoing emergency surgery.
* Patients with an intra aortic balloon pump.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
cerebral oxygen saturation | during surgery

SECONDARY OUTCOMES:
hemodynamic parameters | during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alain Deschamps, MD FRCPC, Principal Investigator — Université de Montréal
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Background] Oberg PA, Sjostrand U. Studies of blood-pressure regulation. I. Common-carotid-artery clamping in studies of the carotid-sinus baroreceptor control of the systemic blood pressure. Acta Physiol Scand. 1969 Mar;75(3):276-86. doi: 10.1111/j.1748-1716.1969.tb04381.x. No abstract available. PMID 5790220
- [Background] Heijman K, Heijman L, Jonzon A, Sedin G, Sjostrand U, Widman B. High frequency positive pressure ventilation during anaesthesia and routine surgery in man. Acta Anaesthesiol Scand. 1972;16(3):176-87. doi: 10.1111/j.1399-6576.1972.tb00588.x. No abstract available. PMID 4566465
- [Background] Ratzenhofer-Komenda B, Prause G, Offner A, Smolle-Juttner FM. Intraoperative application of high frequency ventilation in thoracic surgery. Acta Anaesthesiol Scand Suppl. 1996;109:149-53. No abstract available. PMID 8901989
- [Background] Babinski MF, Smith RB. High frequency ventilation. Int Anesthesiol Clin. 1986 Spring;24(1):75-92. doi: 10.1097/00004311-198602410-00008. No abstract available. PMID 3512455
- [Background] Glenski JA, Crawford M, Rehder K. High-frequency, small-volume ventilation during thoracic surgery. Anesthesiology. 1986 Feb;64(2):211-4. doi: 10.1097/00000542-198602000-00014. PMID 3511770
- [Background] Gallagher TJ, Klain MM, Carlon GC. Present status of high frequency ventilation. Crit Care Med. 1982 Sep;10(9):613-7. doi: 10.1097/00003246-198209000-00013. No abstract available. PMID 7049574
- [Background] Rouby JJ, Simonneau G, Benhamou D, Sartene R, Sardnal F, Deriaz H, Duroux P, Viars P. Factors influencing pulmonary volumes and CO2 elimination during high-frequency jet ventilation. Anesthesiology. 1985 Nov;63(5):473-82. doi: 10.1097/00000542-198511000-00002. PMID 3931506
- [Background] Heres EK, Shulman MS, Krenis LJ, Moon R. High-frequency ventilation with a conventional anesthetic ventilator during cardiac surgery. J Cardiothorac Vasc Anesth. 1995 Feb;9(1):63-5. doi: 10.1016/s1053-0770(05)80057-6. No abstract available. PMID 7718756
- [Background] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242
- [Background] Kadoi Y, Kawahara F, Saito S, Morita T, Kunimoto F, Goto F, Fujita N. Effects of hypothermic and normothermic cardiopulmonary bypass on brain oxygenation. Ann Thorac Surg. 1999 Jul;68(1):34-9. doi: 10.1016/s0003-4975(99)00306-9. PMID 10421111
- [Background] Ueno T, Ikeda K, Matsuyama S. Characteristic changes in cerebral perfusion during on-pump and off-pump coronary artery surgery. Jpn J Thorac Cardiovasc Surg. 2005 Mar;53(3):138-42. doi: 10.1007/s11748-005-0019-5. PMID 15828293
- [Background] Tuman KJ, McCarthy RJ, March RJ, Najafi H, Ivankovich AD. Morbidity and duration of ICU stay after cardiac surgery. A model for preoperative risk assessment. Chest. 1992 Jul;102(1):36-44. doi: 10.1378/chest.102.1.36. PMID 1623792
- [Background] Reich DL, Bodian CA, Krol M, Kuroda M, Osinski T, Thys DM. Intraoperative hemodynamic predictors of mortality, stroke, and myocardial infarction after coronary artery bypass surgery. Anesth Analg. 1999 Oct;89(4):814-22. doi: 10.1097/00000539-199910000-00002. PMID 10512249
- [Background] Tremblay NA, Hardy JF, Perrault J, Carrier M. A simple classification of the risk in cardiac surgery: the first decade. Can J Anaesth. 1993 Feb;40(2):103-11. doi: 10.1007/BF03011305. PMID 8443847
- [Background] Deschamps A, Kaufman I, Backman SB, Plourde G. Autonomic nervous system response to epidural analgesia in laboring patients by wavelet transform of heart rate and blood pressure variability. Anesthesiology. 2004 Jul;101(1):21-7. doi: 10.1097/00000542-200407000-00006. PMID 15220767
- [Background] Malouf JF, Enriquez-Sarano M, Pellikka PA, Oh JK, Bailey KR, Chandrasekaran K, Mullany CJ, Tajik AJ. Severe pulmonary hypertension in patients with severe aortic valve stenosis: clinical profile and prognostic implications. J Am Coll Cardiol. 2002 Aug 21;40(4):789-95. doi: 10.1016/s0735-1097(02)02002-8. PMID 12204512
- [Background] Mishra M, Chauhan R, Sharma KK, Dhar A, Bhise M, Dhole S, Omar A, Kasliwal RR, Trehan N. Real-time intraoperative transesophageal echocardiography--how useful? Experience of 5,016 cases. J Cardiothorac Vasc Anesth. 1998 Dec;12(6):625-32. doi: 10.1016/s1053-0770(98)90232-4. PMID 9854658
- [Background] Bezold LI, Pignatelli R, Altman CA, Feltes TF, Gajarski RJ, Vick GW 3rd, Ayres NA. Intraoperative transesophageal echocardiography in congenital heart surgery. The Texas Children's Hospital experience. Tex Heart Inst J. 1996;23(2):108-15. No abstract available. PMID 8792541
- [Background] Komukai K, Shibata T, Mochizuki S. C-reactive protein is related to impaired oxygenation in patients with acute aortic dissection. Int Heart J. 2005 Sep;46(5):795-9. doi: 10.1536/ihj.46.795. PMID 16272770
- [Background] Puls A, Pollok-Kopp B, Wrigge H, Quintel M, Neumann P. Effects of a single-lung recruitment maneuver on the systemic release of inflammatory mediators. Intensive Care Med. 2006 Jul;32(7):1080-5. doi: 10.1007/s00134-006-0174-x. Epub 2006 May 9. PMID 16791672
- [Background] Tillett WS, Francis Jr T (1930).
- [Background] Lau DC, Dhillon B, Yan H, Szmitko PE, Verma S. Adipokines: molecular links between obesity and atheroslcerosis. Am J Physiol Heart Circ Physiol. 2005 May;288(5):H2031-41. doi: 10.1152/ajpheart.01058.2004. Epub 2005 Jan 14. PMID 15653761
- [Background] Chin KM, Channick RN, Kim NH, Rubin LJ. Central venous blood oxygen saturation monitoring in patients with chronic pulmonary arterial hypertension treated with continuous IV epoprostenol: correlation with measurements of hemodynamics and plasma brain natriuretic peptide levels. Chest. 2007 Sep;132(3):786-92. doi: 10.1378/chest.07-0694. Epub 2007 Jul 23. PMID 17646224
- [Background] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782
- [Background] Denault AY, Couture P, Buithieu J, Haddad F, Carrier M, Babin D, Levesque S, Tardif JC. Left and right ventricular diastolic dysfunction as predictors of difficult separation from cardiopulmonary bypass. Can J Anaesth. 2006 Oct;53(10):1020-9. doi: 10.1007/BF03022532. PMID 16987858
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Pichot V, Gaspoz JM, Molliex S, Antoniadis A, Busso T, Roche F, Costes F, Quintin L, Lacour JR, Barthelemy JC. Wavelet transform to quantify heart rate variability and to assess its instantaneous changes. J Appl Physiol (1985). 1999 Mar;86(3):1081-91. doi: 10.1152/jappl.1999.86.3.1081. PMID 10066727
- [Background] European Cardiovascular disease 2006 - 1-4, NT BNP in stable coronary artery diease
- [Background] Dumesnil JG, Pibarot P. Prosthesis-patient mismatch and clinical outcomes: the evidence continues to accumulate. J Thorac Cardiovasc Surg. 2006 May;131(5):952-5. doi: 10.1016/j.jtcvs.2005.12.032. No abstract available. PMID 16678574
- [Background] Chee TS, Quek SS, Ding ZP, Chua SM. Clinical utility, safety, acceptability and complications of transoesophageal echocardiography (TEE) in 901 patients. Singapore Med J. 1995 Oct;36(5):479-83. PMID 8882528
- [Background] Khoury AF, Afridi I, Quinones MA, Zoghbi WA. Transesophageal echocardiography in critically ill patients: feasibility, safety, and impact on management. Am Heart J. 1994 May;127(5):1363-71. doi: 10.1016/0002-8703(94)90057-4. PMID 8172066
- [Background] Haddad F, Denault AY, Couture P, Cartier R, Pellerin M, Levesque S, Lambert J, Tardif JC. Right ventricular myocardial performance index predicts perioperative mortality or circulatory failure in high-risk valvular surgery. J Am Soc Echocardiogr. 2007 Sep;20(9):1065-72. doi: 10.1016/j.echo.2007.02.017. Epub 2007 Jun 12. PMID 17566702